CLINICAL TRIAL: NCT01136291
Title: Physical Exercise Influence on Maternal, Perinatal Outcomes and Quality of Life Among Overweight and Obese Pregnant Women:
Brief Title: Physical Exercise Influence Among Overweight and Obese Pregnant Women
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Campinas, Brazil (Other)
Responsible Party: University of Campinas, Departamento de tocoginecologia
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: exerciseobesitypregnancy
Record Dates: First submitted 2010-05-21; First posted 2010-06-03 (Estimated); Results first posted 2011-02-23 (Estimated); Last update posted 2011-03-23 (Estimated); Status verified 2011-03

CONDITIONS: Obesity; Overweight
Keywords: pregnancy; obesity; physical exercise; quality of life
MeSH Terms: conditions — Obesity; Overweight; Motor Activity | interventions — Exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- physical exercise (Other): exercise on obese and overweight pregnant women, routine prenatal care and nutritional counseling
  Interventions: Other: physical exercise
- no exercise (No Intervention): Routine prenatal care and nutritional counseling. No exercise

INTERVENTIONS:
Other: physical exercise — The exercise protocol was done under supervision once a week. Pregnant women have been told to do some exercise three more times during the week unsupervised and may be the protocol of exercises or walk in mild to moderate intensity.
  The exercise protocol lasted 50 minutes with 10 minutes of stretching overall, 30 minutes of exercise for muscle strengthening and 10 minutes of relaxation.
  These women also received nutrition counseling and prenatal care.
  Arms: physical exercise

SUMMARY:
Objective: To evaluate the association between physical exercise for obese or overweight women and the maternal, perinatal outcomes and perception of these women about their quality of life.

Methods: A randomized controlled clinical trial with 78 pregnant women. Overweight or obese (BMI ≥ 26 kg / m²), gestational age between 14 and 24 weeks and from age 18 years were included. They will be divided into two random groups: one which will an exercise program under supervision and guidance received from home exercises (study group) and another that followed the standard routine prenatal care service (control group). Both groups will receive standardized nutritional counseling by the department of nutrition and dietetics and a questionnaire measuring quality of life WHOQOL-short at 14 - 24 weeks and at 36 weeks of pregnancy. The intervention results will be analyzed by intention to treat. A P value less than 0.05 will be used to determine statistical significance.

DETAILED DESCRIPTION:
Objective: To evaluate the association between physical exercise for obese or overweight women and the maternal, perinatal outcomes and perception of these women about their quality of life.

Methods: A randomized controlled clinical trial with 78 pregnant women. Overweight or obese (BMI ≥ 26 kg / m²), gestational age between 14 and 24 weeks and from age 18 years were included. They will be divided into two random groups: one which will an exercise program under supervision and guidance received from home exercises (study group) and another that followed the standard routine prenatal care service (control group). Both groups will receive standardized nutritional counseling by the department of nutrition and dietetics and a questionnaire measuring quality of life WHOQOL-short at 14 - 24 weeks and at 36 weeks of pregnancy. The intervention results will be analyzed by intention to treat. A P value less than 0.05 will be used to determine statistical significance.

ELIGIBILITY:
* Overweight or obese (BMI ≥ 26 kg / m²),
* Gestational age between 14 and 24 weeks and from age 18 years
* No contraindication for physical exercise on pregnancy

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 82 (Actual)
Dates: Start 2008-08; Primary Completion 2010-08 (Actual); Study Completion 2010-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Fernanda Surita, MD, PhD, Principal Investigator — University of Campinas, Brazil
Locations (2):
- Brazil (2):
  - Centro de Atenção Integral à saúde da mulher, Campinas, São Paulo
  - Centro de atenção integral à saúde da mulher - CAISM, Campinas, São Paulo

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A randomized controlled clinical trial was conducted with pregnant women seen at the Prenatal Outpatient Clinic of the Women's Integral Healthcare Center (CAISM-UNICAMP) from August 2008 to August 2010.
Pre-assignment Details: The entire study protocol was explained to these women and a written informed consent term was obtained. Subsequently, the women were randomly assigned to two groups: 1) one exercised under supervision and received home exercise counseling (study group) and 2) the other followed the prenatal routine of the service (control group).
Groups:
- Physical Exercise: The exercise protocol was done under supervision once a week. Pregnant women have been told to do some exercise three more times during the week unsupervised and may be the protocol of exercises or walk in mild to moderate intensity.
  The exercise protocol lasted 50 minutes with 10 minutes of stretching overall, 30 minutes of exercise for muscle strengthening and 10 minutes of relaxation.
  These women also received nutrition and prenatal care.
- no Exercise: The pregnant women in this group underwent routine prenatal. In addition to receiving nutritional counseling.
Period: Overall Study
Arm/Group | Physical Exercise | no Exercise
Started | 40 | 42
Follow | 40 | 42
Completed | 39 | 41
Not Completed | 1 | 1
Not completed — Lost to Follow-up | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Physical Exercise | no Exercise | Total
Number analyzed (Participants) | 40 | 42 | 82
Age Continuous [Mean (Standard Deviation); unit: years] | 29.7 (6.8) | 30.9 (5.9) | 30.1 (6.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 40 | 42 | 82
  Male | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  Brazil | 40 | 42 | 82

OUTCOME MEASURES:

1. Primary Outcome: Gestational Weight Gain
Description: Gestational weight gain is the difference between the prepregnancy weight and the last weight measure at the end of pregnancy
Time Frame: baseline and at 40 gestational weeks
Measure: Mean (Standard Deviation); unit: kg
Arm/Group | Physical Exercise | no Exercise
Number analyzed (Participants) | 40 | 42
kg | 10.3 (5.0) | 11.5 (7.4)
Statistical Analysis 1: Comparison: Physical Exercise vs no Exercise; The homogeneity between the groups was compared by the Student's t test or the Mann-Whitney test for continuous variables and chi-square for categorical variables.A comparison between values before and after the study group session was performed by the Student's t test. The effect of the exercise was evaluated by repeated measures ANOVA, where the effect of time and group were evaluated on pressure, weight, Body Mass Index (BMI)and World Health Organization Quality of Life Questionnarie domains; Test type: Superiority or Other; p < 0.05, t-test, 1 sided

2. Primary Outcome: Weight Gain During the Program
Description: Weight gain during the program was the difference between the weight measured at study entry and final consultation weight, measured by a mechanical scale, in kilos and grams
Time Frame: at the 14 to 40 gestational weeks
Measure: Mean (Standard Deviation); unit: kg
Arm/Group | Physical Exercise | no Exercise
Number analyzed (Participants) | 40 | 42
kg | 7.7 (4.3) | 8.1 (4.3)

3. Secondary Outcome: Quality of Life Through World Health Organization Quality of Life Abbreviated Questionnaire WHOQOL-Bref)
Description: All pregnant women responded to the quality of life WHOQOL-bref questionnaire, at study inclusion and at the completion of 36 gestational weeks. The domains of these questionnaires were calculated on a scale of zero (the worse quality of life) to 100 points (the better quality of life).
Time Frame: at the 14 and at the 40 gestational weeks
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Physical Exercise | no Exercise
Number analyzed (Participants) | 40 | 42
scores on a scale | 49.8 (17.1) | 42.2 (16.1)

ADVERSE EVENTS:
Arm/Group | Physical Exercise | no Exercise
Serious Adverse Events (participants affected / at risk) | 0/40 | 0/42
Other Adverse Events (participants affected / at risk) | 0/40 | 0/42

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No